CLINICAL TRIAL: NCT03105310
Title: Pegylated Interferon Alone or in Combination With Ezetimibe for Patients With Chronic Hepatitis D
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Zaigham Abbas, Consultant Gastroenterologist, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3636-Med-ERC
Record Dates: First submitted 2017-03-26; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis D, Chronic
Keywords: Hepatitis D; Ezetimibe; Pegylated interferon
MeSH Terms: conditions — Hepatitis D, Chronic; Hepatitis D | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pegylated interferon (Active Comparator): Pegylated interferon alfa alone 180 microgram subcutaneous weekly for 24 weeks
  Interventions: Drug: Pegylated interferon alfa
- Pegylated interferon with ezetimibe (Experimental): Pegylated interferon alfa 180 micro-gram subcutaneous weekly for 24 weeks and Ezetimibe 10 mg orally for 24 weeks
  Interventions: Drug: Pegylated interferon alfa; Drug: Ezetimibe

INTERVENTIONS:
Drug: Pegylated interferon alfa — Pegylated interferon alfa
Drug: Ezetimibe — Ezetimibe
  Arms: Pegylated interferon with ezetimibe

SUMMARY:
Ezetimibe possesses pharmacophore features to inhibit NTCP, the receptor required for HBV and HDV hepatocyte entry, that include two hydrophobes and one hydrogen bond acceptor.

The aim of the study io evaluate the utility of Ezetimibe in combination with pegylated interferon in patients with chronic HDV infection.

ELIGIBILITY:
Inclusion Criteria:

* Presence of anti-HDV in serum
* Presence of quantifiable HDV RNA in serum
* Elevated ALT > ULN

Exclusion Criteria:

* Decompensated liver disease
* Patients with ALT levels greater than 10 times ULN (400 U/L)
* Pregnancy or inability to practice adequate contraception.
* Significant systemic or major illnesses other than liver disease, including, but not limited to, congestive heart failure, renal failure (eGFR <50 ml/min), organ transplantation, serious psychiatric disease or depression and active coronary artery disease.
* Systemic immunosuppressive therapy
* Evidence of another form of liver disease in addition to viral hepatitis
* Active substance abuse, such as alcohol or injection drugs
* Hepatocellular carcinoma
* Concurrent hepatitis C infection or HIV coinfection
* Diagnosis of malignancy in the five years
* Concurrent usage of statins
* Concurrent use of any other drug known to inhibit NTCP
* Inability to understand or sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in HDV RNA quantitative measurements of >2 logs from baseline | 24 weeks of therapy

IPD SHARING:
Plan to Share IPD: No